CLINICAL TRIAL: NCT00896363
Title: A Randomised, Double-Blind, Parallel-Group, Placebo-Controlled Study Evaluating the Efficacy and Safety of GSK163090 in Subjects With Major Depressive Disorder
Brief Title: Safety and Efficacy Study in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 109035
Record Dates: First submitted 2009-05-07; First posted 2009-05-11 (Estimated); Results first posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2017-08

CONDITIONS: Depressive Disorder
Keywords: anti-depressant; Severe Depression; Efficacy; Major Depressive Disorder; Major Depressive Episode
MeSH Terms: conditions — Depressive Disorder; Depression; Depressive Disorder, Major | interventions — 1-(3-(2-(4-(2-methyl-5-quinolinyl)-1-piperazinyl)ethyl)phenyl)-2-imidazolidinone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Active Comparator): Parallel Group - High Dose Arm, Low Dose Arm
  Interventions: Drug: GSK163090 1 mg; Drug: GSK163090 3 mg
- Placebo (Placebo Comparator): Parallel Group
  Interventions: Drug: GSK163090 Placebo

INTERVENTIONS:
Drug: GSK163090 1 mg — Developed for the treatment of Major Depressive Disorder
  Arms: Active
Drug: GSK163090 Placebo — Developed for the treatment of Major Depressive Disorder
  Arms: Placebo
Drug: GSK163090 3 mg — Developed for the treatment of Major Depressive Disorder
  Arms: Active

SUMMARY:
The purpose of this study is to test if GSK163090 can reduce the symptoms of depression. The safety and how well the body can handle the drug will also be investigated. The study will be conducted in Russia in hospitalised patients with severe depression. GSK163090 will be compared with placebo, which looks like the study drug but does not contain any active substance. Subjects will be given either the study drug or the matching placebo.

DETAILED DESCRIPTION:
This is a randomised, multi-centre, double-blind, placebo-controlled, repeat dose, parallel group study in male and female patients with severe depression requiring hospitalization. Efficacy, safety and tolerability will be assessed in three treatment arms. The study will consist of a screening period, a treatment phase (up to 6 weeks) and a post-treatment follow-up visit. The study duration from screening to follow up will be approximately 9 weeks. Subjects who pass screening will be randomized on Day 1 to one of three treatment arms (low dose arm, high dose arm or placebo). Each treatment arm will contain approximately 50 subjects. The subject's depressive symptoms will be assessed using the HAMD17- CR.

ELIGIBILITY:
Inclusion Criteria:

* Currently have severe depression (Major Depressive Disorder - without psychotic features)
* meet criteria (DSM IV-TR ) for current major depressive episode for at least 4 weeks but for no greater than 24 months
* depression questionnaire (HAMD17) total score greater than or equal to 24
* subject must read and able to give written informed consent
* male or female 18 to 64 years
* use appropriate birth control method
* BMI 18.8 - 35.0 kg/m2 (inclusive)

Exclusion Criteria:

* Primary diagnosis of other psychiatric disorders
* thoughts of killing ones self or someone else
* taking psychiatric medicine or therapy within the six months
* Has previously failed an adequate course of medication for MDD from two different classes of antidepressants.
* Unstable medical disorder or a disorder that would interfere with the action of the drug
* Abuse of alcohol or drugs
* Past history of serotonin syndrome or a history of clinical significant intolerance of SSRIs (class of drugs used for depression).
* History of migraine headaches that respond to treatment with triptan medication.
* History of a clinically significant abnormality of the neurological system (including dementia and other cognitive disorders or significant head injury) or any history of seizure (excluding febrile seizure).
* Currently taking part in another clinical study or has done so within six months
* Pregnant, planning to become pregnant shortly or breastfeeding
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2009-04-23 (Actual); Primary Completion 2010-02-09 (Actual); Study Completion 2010-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- Russia (9):
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Lipetsk Region
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 109035 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109035 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109035 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 109035 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109035 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109035 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 109035 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 99 participants with major depressive disorder (MDD) were enrolled in this study. The study was conducted at sixteen centers in Russia from 23 April 2009 to 09 February 2010
Groups:
- Placebo: Participants were randomized to receive oral dose of matching placebo tablet to GSK163090 twice a day, with one tablet in the morning (AM) and one taken between 11 to 13 hours after the AM dose in the evening (PM) for 6 weeks.
- GSK163090 1 mg: Participants were randomized to the low dose arm to receive oral dose of GSK163090 up to 1 milligram (mg) immediate release tablet twice a day, with one tablet in the AM and one taken between 11 to 13 hours after the AM dose in the PM for 6 weeks. Daily dosage was provided according to the titration schedule, where the participants received (AM -matching placebo tablet, PM- GSK163090 0.5 mg ) on Day 1 and continued (AM- GSK163090 0.5 mg and PM- GSK163090 0.5 mg) from Day 2 onwards
- GSK163090 3 mg: Participants were randomized to the high dose arm to receive oral dose of GSK163090 up to 3 mg immediate release tablet twice a day, with one tablet in the AM and one taken between 11 to 13 hours after the AM dose in the PM for 6 weeks. Daily dosage was provided according to the titration schedule, where the participants received (AM -matching placebo tablet, PM- GSK163090 0.5 mg ) on Day 1, (AM- GSK163090 0.5 mg and PM- GSK163090 0.5 mg) on Day 2 to Day 3, (AM- GSK163090 1 mg and PM- GSK163090 1 mg) on Day 4 to Day 5 and continued (AM- GSK163090 1.5 mg and PM- GSK163090 1.5 mg) from Day 6 onwards.
Period: Overall Study
Arm/Group | Placebo | GSK163090 1 mg | GSK163090 3 mg
Started | 31 | 36 | 32
Completed | 25 | 25 | 24
Not Completed | 6 | 11 | 8
Not completed — Adverse Event | 3 | 4 | 2
Not completed — Lack of Efficacy | 0 | 2 | 1
Not completed — Withdrawal by Subject | 3 | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants were randomized to receive oral dose of matching placebo tablet to GSK163090 twice a day, with one tablet AM and one taken between 11 to 13 hours after the AM dose in the PM for 6 weeks.
- GSK163090 1 mg: Participants were randomized to the low dose arm to receive oral dose of GSK163090 up to 1 mg immediate release tablet twice a day, with one tablet in the AM and one taken between 11 to 13 hours after the AM dose in the PM for 6 weeks. Daily dosage was provided according to the titration schedule, where the participants received (AM -matching placebo tablet, PM- GSK163090 0.5 mg ) on Day 1 and continued (AM- GSK163090 0.5 mg and PM- GSK163090 0.5 mg) from Day 2 onwards.
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK163090 1 mg | GSK163090 3 mg | Total
Number analyzed (Participants) | 31 | 36 | 32 | 99
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.7 (11.12) | 42.2 (14.57) | 47.3 (10.84) | 43.4 (12.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 21 | 62
  Male | 11 | 15 | 11 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 30 | 36 | 32 | 98
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Hamilton Depression Rating Scale (HAMD17), on Day 14 and 42
Description: HAMD-17 is a 17-item scale that evaluates depressed mood, vegetative and cognitive symptoms of depression, and co-morbid anxiety symptoms. The 17 items were rated on either a 5-point (0-4) or a 3-point (0-2) scale. In general, the 5 point scale items use a rating of 0=absent; 1=doubtful to mild; 2=mild to moderate; 3=moderate to severe; 4=very severe. The 3-point scale items use a rating of 0=absent; 1=probable or mild; 2=definite. The total HAMD-17score ranges from 0 (not ill) to 52 (severely ill). The highest possible score was 52, which represented the most severe measure of depression; the lowest possible score was 0, which represents an absence of depression. Baseline was defined as the assessment done on Day 1 (pre-dose). Change from baseline in total Score was the difference between HAMD total score at the time point being analyzed to Day 1.
Time Frame: Baseline (Day 1, pre-dose), Day 14 and Day 42
Population: Intent-to-treat population comprised of all participants who gave informed consent, were randomized, received at least one dose of double blind medication and for whom at least one post-randomization assessment was available. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | GSK163090 1 mg | GSK163090 3 mg
Number analyzed (Participants) | 31 | 36 | 32
Score on scale
  DAY 14: number analyzed (Participants) | 28 | 34 | 29
  DAY 14 | -10.9 (6.02) | -10.8 (5.68) | -10.3 (5.95)
  DAY 42: number analyzed (Participants) | 25 | 25 | 26
  DAY 42 | -18.6 (8.21) | -18.4 (6.54) | -16.7 (8.11)
Statistical Analysis 1: Comparison: Placebo vs GSK163090 1 mg; Comparison of placebo and GSK163090 1 mg on Day 14; Test type: Superiority or Other; Mixed model repeated measures analysis; Mean Difference (Net) = 0.85, 90% CI 2-sided [-1.62 to 3.32] — The point estimate was calculated as least square mean difference (net values) of HAMD17
Statistical Analysis 2: Comparison: Placebo vs GSK163090 3 mg; Comparison of placebo and GSK163090 3 mg on Day 14; Test type: Superiority or Other; Mixed model repeated measures analysis; Mean Difference (Net) = 0.33, 90% CI 2-sided [-2.12 to 2.78] — The point estimate was calculated as least square mean difference (net values) of HAMD17
Statistical Analysis 3: Comparison: Placebo vs GSK163090 1 mg; Comparison of placebo and GSK163090 1 mg on Day 42; Test type: Superiority or Other; Mixed model repeated measures analysis; Mean Difference (Net) = 1.57, 90% CI 2-sided [-2.01 to 5.14] — The point estimate was calculated as least square mean difference (net values) of HAMD17
Statistical Analysis 4: Comparison: Placebo vs GSK163090 3 mg; Comparison of placebo and GSK163090 3 mg on Day 42; Test type: Superiority or Other; Mixed model repeated measures analysis; Mean Difference (Net) = 1.66, 90% CI 2-sided [-1.81 to 5.13] — The point estimate was calculated as least square mean difference (net values) of HAMD17

2. Primary Outcome: Change From Baseline in Bech Melancholia Subscale (BECH 6) Scale, on Day 14 and 42
Description: The bech melancholia is sum of scores on 6 items- depressed mood, feelings of guilt, work and activities, retardation, anxiety psychic, somatic symptoms general (items 1, 2, 7, 8, 10 and 13 respectively). Each item having 5 responses. The items are rated on a scale of 0-4, where 0=absent; 1=doubtful to mild; 2=mild to moderate; 3=moderate to severe; 4=very severe. Total possible score is 0-24. where the lowest possible score was 0, which represented an absence of depression and higher scores reflecting greater severity of diseases. Baseline was defined as the assessment done on Day 1. Change from baseline was the difference between BECH 6 scale at the time point being analyzed to randomization.
Time Frame: Baseline (Day 1, pre-dose), Day 14 and Day 42
Population: Intent-to-treat population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | GSK163090 1 mg | GSK163090 3 mg
Number analyzed (Participants) | 31 | 36 | 32
Score on scale
  DAY 14: number analyzed (Participants) | 28 | 34 | 29
  DAY 14 | -4.9 (3.14) | -4.6 (2.85) | -4.2 (3.33)
  DAY 42: number analyzed (Participants) | 25 | 25 | 26
  DAY 42 | -8.7 (4.19) | -8.4 (3.30) | -7.8 (4.36)
Statistical Analysis 1: Comparison: Placebo vs GSK163090 1 mg; Comparison of placebo and GSK163090 1 mg on Day 14; Test type: Superiority or Other; Mixed model repeated measures analysis; Mean Difference (Net) = 0.31, 90% CI 2-sided [-0.93 to 1.56] — The point estimate was calculated as least square mean difference (net values) of BECH 6 scale
Statistical Analysis 2: Comparison: Placebo vs GSK163090 3 mg; Comparison of placebo and GSK163090 3 mg on Day 14; Test type: Superiority or Other; Mixed model repeated measures analysis; Mean Difference (Net) = 0.51, 90% CI 2-sided [-0.73 to 1.75] — The point estimate was calculated as least square mean difference (net values) of BECH 6 scale
Statistical Analysis 3: Comparison: Placebo vs GSK163090 1 mg; Comparison of placebo and GSK163090 1 mg on Day 42; Test type: Superiority or Other; Mixed model repeated measures analysis; Mean Difference (Net) = 0.66, 90% CI 2-sided [-1.10 to 2.42] — The point estimate was calculated as least square mean difference (net values) of BECH 6 scale
Statistical Analysis 4: Comparison: Placebo vs GSK163090 3 mg; Comparison of placebo and GSK163090 3 mg on Day 42; Test type: Superiority or Other; Mixed model repeated measures analysis; Mean Difference (Net) = 0.77, 90% CI 2-sided [-0.93 to 2.48] — The point estimate was calculated as least square mean difference (net values) of BECH 6 scale

3. Primary Outcome: Change From Baseline in Quick Inventory of Depressive Symtomatology - Self Rated (QIDS-SR) Scale, on Day 14 and 42
Description: The QIDS-SR is a 16-item, participant-rated short form of the Inventory of Depressive Symptomatology that assesses 9 domains: sad mood, concentration, self-criticism, suicidal ideation, interest, energy/fatigue, sleep disturbance (initial, middle, and late insomnia or hypersomnia), appetite/weight increase/decrease and psychomotor agitation/retardation. A total score was obtained by summing scores on each domain. the scores ranges from 0 (none) to 27 (very severe), where the highest possible score was 27, which represented the most severe measure of depression; the lowest possible score was 0, which represents an absence of depression. Baseline was defined as the assessment done on Day 1. Change from Randomization in total score was the difference between QIDS total score at the time point being analyzed to randomization.
Time Frame: Baseline (Day 1, pre-dose), Day 14 and Day 42
Population: Intent-to-treat population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | GSK163090 1 mg | GSK163090 3 mg
Number analyzed (Participants) | 31 | 36 | 32
Score on scale
  Day 14: number analyzed (Participants) | 28 | 34 | 28
  Day 14 | -6.2 (3.40) | -6.1 (4.19) | -6.5 (3.96)
  DAY 42: number analyzed (Participants) | 20 | 24 | 24
  DAY 42 | -11.0 (4.75) | -11.4 (4.32) | -10.8 (4.57)
Statistical Analysis 1: Comparison: Placebo vs GSK163090 1 mg; Comparison of placebo and GSK163090 1 mg on Day 14; Test type: Superiority or Other; Mixed model repeated measures analysis; Mean Difference (Net) = 0.72, 90% CI 2-sided [-0.94 to 2.37] — The point estimate was calculated as least square mean difference (net values) of QIDS-SR scale
Statistical Analysis 2: Comparison: Placebo vs GSK163090 3 mg; Comparison of placebo and GSK163090 3 mg on Day 14; Test type: Superiority or Other; Mixed model repeated measures analysis; Mean Difference (Net) = -0.44, 90% CI 2-sided [-2.10 to 1.21] — The point estimate was calculated as least square mean difference (net values) of QIDS-SR scale
Statistical Analysis 3: Comparison: Placebo vs GSK163090 1 mg; Comparison of placebo and GSK163090 1 mg on Day 42; Test type: Superiority or Other; Mixed model repeated measures analysis; Mean Difference (Net) = 0.84, 90% CI 2-sided [-1.22 to 2.90] — The point estimate was calculated as least square mean difference (net values) of QIDS-SR scale
Statistical Analysis 4: Comparison: Placebo vs GSK163090 3 mg; Comparison of placebo and GSK163090 3 mg on Day 42; Test type: Superiority or Other; Mixed model repeated measures analysis; Mean Difference (Net) = 0.81, 90% CI 2-sided [-1.22 to 2.85] — The point estimate was calculated as least square mean difference (net values) of QIDS-SR scale

4. Primary Outcome: Number of Participants With Suicidal Behavior and Suicidal Ideation Subscales of the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS was a clinician-rated scale that evaluated severity and change of suicidality by integrating both behaviour and ideation. The 2 of 3 sections of the scale were suicidal behavior and suicidal ideation. For suicidal behaviour participants were scored as non-suicidal-0, preparatory acts or behavior communicating ideation-01, aborted attempt-2, interrupted attempt-3 or actual attempt-4. The score ranges from 0-4, where 0 was absence of suicidal behavior and 4 being the most severe form of suicidal behavior. On the Suicidal Ideation scale, participants were scored as non-suicidal-0, wish to be dead-1, non-specific active suicidal thoughts-2, active suicidal ideation with associated thoughts of methods without intent-3, active suicidal ideation with some intent to act on suicidal thoughts without clear plan-4, active suicidal ideation with plan and intent-5. The score ranges from 0-5, where 0 was absence of suicidal ideation and 5 being the most severe form of suicidal ideation.
Time Frame: Up to Day 52
Population: All subjects population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK163090 1 mg | GSK163090 3 mg
Number analyzed (Participants) | 31 | 36 | 32
Participants
  suicidal behavior | 0 | 0 | 0
  suicidal ideation,Day1,Wish to be dead | 7 | 5 | 4
  suicidal ideation,Day14,Wish to be dead | 1 | 1 | 1

5. Primary Outcome: Number of Participants With Abnormal Hematology Values of Clinical Concern Range (CCR).
Description: Only those parameters for which at least one value of CC was reported were summarized. Pre-defined limits of CC (CC Low [relative to the lower limit of normal], CC High [relative to the upper limit of normal]) were: hemoglobin (Hb): > 25, 180; hematocrit (Hct): > 0.075, 0.54; absolute neutrophil count (ANC): < 1.5, NA; platelet: < 100, > 550; white blood cells (WBC): < 3,> 20
Time Frame: Up to Day 42
Population: All subjects population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK163090 1 mg | GSK163090 3 mg
Number analyzed (Participants) | 31 | 36 | 32
Participants
  Hb,screening, Low: number analyzed (Participants) | 28 | 35 | 30
  Hb,screening, Low | 2 | 0 | 0
  Hb,Day 14, Low: number analyzed (Participants) | 24 | 31 | 23
  Hb,Day 14, Low | 2 | 0 | 0
  Hct,screening, Low: number analyzed (Participants) | 28 | 35 | 30
  Hct,screening, Low | 2 | 0 | 0
  ANC,screening, Low: number analyzed (Participants) | 28 | 35 | 30
  ANC,screening, Low | 1 | 0 | 0
  ANC,Day14, Low: number analyzed (Participants) | 24 | 31 | 23
  ANC,Day14, Low | 1 | 1 | 1
  ANC,Day42, Low: number analyzed (Participants) | 22 | 23 | 23
  ANC,Day42, Low | 1 | 0 | 1
  Platelet,screening, High: number analyzed (Participants) | 28 | 35 | 30
  Platelet,screening, High | 1 | 0 | 0
  Platelet,Day 14, High: number analyzed (Participants) | 24 | 31 | 23
  Platelet,Day 14, High | 1 | 0 | 0
  Platelet,Day 42, High: number analyzed (Participants) | 22 | 23 | 23
  Platelet,Day 42, High | 1 | 0 | 0
  WBC,Day 14, High | 0 | 2 | 0
  WBC,Day 14, Low | 1 | 1 | 1
  WBC,Day 42, Low: number analyzed (Participants) | 22 | 23 | 23
  WBC,Day 42, Low | 1 | 0 | 1

6. Primary Outcome: Number of Participants With Abnormal Chemistry Values of CCR
Description: Only those parameters for which at least one value of CC was reported were summarized. Pre-defined limits of CC (CC Low [relative to the lower limit of normal], CC High [relative to the upper limit of normal]) were: albumin (unit: gram per liter): < 30, NA; alanine aminotransferase (ALT): NA, >= 3 times upper limit of normal; aspartate aminotransferase (AST): NA, >= 3 times upper limit of normal; total bilirubin: NA, >=1.5 times upper limit of normal; calcium: < 2.0, > 2.75; gamma glutamyl transferase (GGT): < 3.0, > 9; potassium: < 3.0, > 5.5; magnesium: < 0.5, > 1.23.
Time Frame: Up to Day 42
Population: All subjects population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK163090 1 mg | GSK163090 3 mg
Number analyzed (Participants) | 31 | 36 | 32
Participants
  Albumin,screening, High: number analyzed (Participants) | 31 | 36 | 30
  Albumin,screening, High | 0 | 1 | 1
  Albumin,Day 14, High: number analyzed (Participants) | 28 | 33 | 28
  Albumin,Day 14, High | 1 | 1 | 0
  ALT,Day 14, High: number analyzed (Participants) | 28 | 33 | 28
  ALT,Day 14, High | 1 | 0 | 0
  ALT,Day 42, High: number analyzed (Participants) | 25 | 24 | 24
  ALT,Day 42, High | 0 | 1 | 0
  AST,Day 42, High: number analyzed (Participants) | 25 | 24 | 24
  AST,Day 42, High | 0 | 1 | 0
  Total bilirubin,screening, High: number analyzed (Participants) | 31 | 36 | 30
  Total bilirubin,screening, High | 0 | 1 | 0
  Total bilirubin,Day 7, High: number analyzed (Participants) | 30 | 35 | 30
  Total bilirubin,Day 7, High | 0 | 1 | 0
  Calcium,Day14, Low: number analyzed (Participants) | 28 | 33 | 28
  Calcium,Day14, Low | 1 | 0 | 1
  GGT,screening, High: number analyzed (Participants) | 31 | 36 | 30
  GGT,screening, High | 1 | 2 | 1
  GGT,Day14, High: number analyzed (Participants) | 28 | 33 | 28
  GGT,Day14, High | 1 | 1 | 1
  GGT,Day42, High: number analyzed (Participants) | 25 | 24 | 24
  GGT,Day42, High | 0 | 2 | 0
  Glucose,screening, High: number analyzed (Participants) | 31 | 36 | 30
  Glucose,screening, High | 1 | 1 | 1
  Glucose,Day 14, High: number analyzed (Participants) | 28 | 33 | 28
  Glucose,Day 14, High | 0 | 4 | 1
  Glucose,Day42, High: number analyzed (Participants) | 25 | 24 | 24
  Glucose,Day42, High | 0 | 2 | 1
  Potassium,Day 14, High: number analyzed (Participants) | 28 | 33 | 28
  Potassium,Day 14, High | 0 | 0 | 1
  Magnesium,screening, High: number analyzed (Participants) | 31 | 36 | 30
  Magnesium,screening, High | 0 | 2 | 0
  Magnesium,Day 14, High: number analyzed (Participants) | 28 | 33 | 28
  Magnesium,Day 14, High | 1 | 0 | 1
  Magnesium,Day 42, High: number analyzed (Participants) | 25 | 24 | 24
  Magnesium,Day 42, High | 0 | 0 | 1

7. Primary Outcome: Change From Baseline in Liver Chemistry -Alkaline Phosphatase (ALP), ALT, AST and GGT
Description: Clinical liver chemistry parameters of Alkaline Phosphatase , ALT, AST, GGT were assessed on screening, Day 7, Day 14, Day 28 and Day 42. Screening was defined as Baseline. Change from Baseline in liver chemistry was the difference between the value at time point analyzed and screening.
Time Frame: Baseline (screening) up to Day 42
Population: All subjects population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International unit per litre (IU/L)
Arm/Group | Placebo | GSK163090 1 mg | GSK163090 3 mg
Number analyzed (Participants) | 31 | 36 | 32
International unit per litre (IU/L)
  ALP,Day7: number analyzed (Participants) | 30 | 34 | 28
  ALP,Day7 | 2.8 (21.57) | -6.6 (25.51) | -1.7 (21.77)
  ALP,Day14: number analyzed (Participants) | 28 | 33 | 26
  ALP,Day14 | 4.6 (32.99) | 2.5 (9.79) | -5.4 (26.57)
  ALP,Day28: number analyzed (Participants) | 27 | 26 | 25
  ALP,Day28 | -2.1 (14.92) | -0.8 (20.47) | 0.8 (13.12)
  ALP,Day42: number analyzed (Participants) | 25 | 24 | 23
  ALP,Day42 | -1.1 (12.57) | 8.7 (45.92) | 0.2 (14.37)
  ALT,Day7: number analyzed (Participants) | 30 | 34 | 28
  ALT,Day7 | -1.0 (14.85) | 0.0 (14.20) | -1.4 (3.86)
  ALT,Day14: number analyzed (Participants) | 28 | 32 | 26
  ALT,Day14 | 7.3 (35.81) | -1.9 (15.96) | -2.8 (5.93)
  ALT,Day28: number analyzed (Participants) | 27 | 26 | 25
  ALT,Day28 | -2.8 (5.97) | -2.9 (13.49) | 0.1 (11.43)
  ALT,Day42: number analyzed (Participants) | 25 | 24 | 23
  ALT,Day42 | -2.7 (10.88) | 34.0 (189.18) | -1.9 (6.68)
  AST,Day7: number analyzed (Participants) | 30 | 35 | 28
  AST,Day7 | -1.3 (9.91) | -1.2 (7.07) | -1.7 (6.83)
  AST,Day14: number analyzed (Participants) | 28 | 33 | 26
  AST,Day14 | 1.8 (15.66) | -2.8 (13.62) | -3.2 (7.96)
  AST,Day28: number analyzed (Participants) | 27 | 26 | 25
  AST,Day28 | -1.6 (4.80) | -3.6 (12.45) | -1.6 (7.93)
  AST,Day42: number analyzed (Participants) | 25 | 24 | 23
  AST,Day42 | -1.8 (5.35) | 31.6 (174.14) | -2.3 (7.54)
  GGT,Day14: number analyzed (Participants) | 28 | 33 | 26
  GGT,Day14 | 11.1 (52.04) | 1.7 (23.67) | -5.2 (18.93)
  GGT,Day42: number analyzed (Participants) | 25 | 24 | 23
  GGT,Day42 | -1.8 (16.22) | 12.7 (75.43) | -8.6 (18.22)

8. Primary Outcome: Change From Baseline in Liver Chemistry- Direct Bilirubin and Total Bilirubin
Description: Liver chemistry parameters: Direct Bilirubin and Total Bilirubin were assessed on screening, Day 7, Day 14, Day 28 and Day 42. Screening was defined as Baseline. Change from Baseline in liver chemistry was the difference between the value at time point analyzed and screening.
Time Frame: Baseline (screening) up to Day 42
Population: All subjects population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: UMOL/L
Arm/Group | Placebo | GSK163090 1 mg | GSK163090 3 mg
Number analyzed (Participants) | 31 | 36 | 32
UMOL/L
  Direct bilirubin,Day 7: number analyzed (Participants) | 30 | 35 | 28
  Direct bilirubin,Day 7 | 0.59 (1.745) | 0.13 (1.511) | 0.38 (1.142)
  Direct bilirubin,Day 14: number analyzed (Participants) | 28 | 33 | 26
  Direct bilirubin,Day 14 | 0.61 (1.490) | -0.14 (1.369) | 0.25 (0.845)
  Direct bilirubin,Day 28: number analyzed (Participants) | 27 | 26 | 25
  Direct bilirubin,Day 28 | 0.66 (1.270) | -0.44 (1.541) | 0.06 (1.227)
  Direct bilirubin,Day 42: number analyzed (Participants) | 25 | 24 | 23
  Direct bilirubin,Day 42 | 0.31 (1.508) | -0.08 (1.517) | 0.43 (0.716)
  Total bilirubin,Day 7: number analyzed (Participants) | 30 | 35 | 28
  Total bilirubin,Day 7 | 1.36 (4.465) | 0.66 (3.536) | 1.05 (3.771)
  Total bilirubin,Day 14: number analyzed (Participants) | 28 | 33 | 26
  Total bilirubin,Day 14 | 1.24 (4.040) | -0.33 (3.696) | 0.59 (2.211)
  Total bilirubin,Day 28: number analyzed (Participants) | 27 | 26 | 25
  Total bilirubin,Day 28 | 1.81 (3.421) | -1.05 (4.218) | 0.33 (3.251)
  Total bilirubin,Day 42: number analyzed (Participants) | 25 | 24 | 23
  Total bilirubin,Day 42 | 0.88 (4.056) | -0.30 (3.610) | 1.28 (2.704)

9. Primary Outcome: Number of Participant of Urinanalysis Assessment Over Period
Description: Urinalysis parameters included: Urine Occult Blood, Urine Ketones, Urine Ketones. data for number of participants with abnormal urinanalysis parameters was reported by dipstick method. dipstick was a strip used to detect the presence or absence of these parameters in the urine sample. dipstick test gives results in a semi-quantitative manner, and results can be read as negative, Trace, 1+, 2+, and 3+, indicating proportional concentrations in the urine sample. Urine occult blood dipstick and urine general dipstick were semi quantitative results. Urine glucose and urine ketones dipstick results were in milimole per liter, urine protein dipstick results were in gram per liter.
Time Frame: Screening (Day -10 to -2), Day 14 and Day 42
Population: All subjects population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK163090 1 mg | GSK163090 3 mg
Number analyzed (Participants) | 31 | 36 | 32
Participants
  screening ,urine Occult Blood,+ | 2 | 2 | 1
  screening ,urine Occult Blood,++ | 4 | 0 | 2
  screening ,urine Occult Blood,+++ | 1 | 3 | 0
  screening,urine General,positive: number analyzed (Participants) | 31 | 36 | 31
  screening,urine General,positive | 10 | 17 | 9
  screening,urine ketones,(1) | 1 | 0 | 0
  screening,urine ketones,(4) | 0 | 1 | 0
  screening,urine protein,(0.1) | 1 | 2 | 5
  screening,urine protein,(0.2) | 2 | 6 | 3
  screening,urine protein, (0.3) | 0 | 2 | 2
  Day 14 ,urine Occult Blood,+: number analyzed (Participants) | 20 | 27 | 16
  Day 14 ,urine Occult Blood,+ | 0 | 1 | 0
  Day 14 ,urine Occult Blood,++: number analyzed (Participants) | 20 | 27 | 16
  Day 14 ,urine Occult Blood,++ | 2 | 0 | 1
  Day 14 ,urine Occult Blood,+++: number analyzed (Participants) | 20 | 27 | 16
  Day 14 ,urine Occult Blood,+++ | 1 | 0 | 0
  Day 14,urine General,positive: number analyzed (Participants) | 20 | 27 | 16
  Day 14,urine General,positive | 8 | 13 | 3
  Day 14,urine protein,(0.1): number analyzed (Participants) | 20 | 27 | 16
  Day 14,urine protein,(0.1) | 3 | 1 | 1
  Day 14,urine protein,(0.2): number analyzed (Participants) | 20 | 27 | 16
  Day 14,urine protein,(0.2) | 0 | 5 | 0
  Day 14,urine protein, (0.3): number analyzed (Participants) | 20 | 27 | 16
  Day 14,urine protein, (0.3) | 1 | 1 | 0
  Day 14,urine protein,(0.5): number analyzed (Participants) | 20 | 27 | 16
  Day 14,urine protein,(0.5) | 1 | 1 | 0
  Day 42,urine occult Blood,+: number analyzed (Participants) | 16 | 21 | 12
  Day 42,urine occult Blood,+ | 1 | 2 | 1
  Day 42,urine occult Blood,++: number analyzed (Participants) | 20 | 27 | 16
  Day 42,urine occult Blood,++ | 1 | 2 | 0
  Day 42,urine general,positive: number analyzed (Participants) | 16 | 21 | 12
  Day 42,urine general,positive | 3 | 9 | 5
  Day 42,urine protein,(0.1): number analyzed (Participants) | 16 | 21 | 12
  Day 42,urine protein,(0.1) | 1 | 5 | 1
  Day 42,urine protein,(0.2): number analyzed (Participants) | 16 | 21 | 12
  Day 42,urine protein,(0.2) | 1 | 0 | 1
  Day 42,urine protein,(0.3): number analyzed (Participants) | 16 | 21 | 12
  Day 42,urine protein,(0.3) | 0 | 1 | 2
  Day 42,urine protein,(0.5): number analyzed (Participants) | 16 | 21 | 12
  Day 42,urine protein,(0.5) | 0 | 1 | 0

10. Primary Outcome: Change From Baseline in Electrocardiogram (ECG) Values -PR Interval, QRS Duration, QT Interval, QTcB, QTcF, RR Interval
Description: Data for change from Baseline was reported for PR Interval, QRS Duration, QT Interval, QTcB, QTcF, and RR Interval. 12-lead ECGs was obtained at each time point during the study using an ECG machine that automatically calculated the heart rate and measures PR, QRS, QT, and QTcB ,QTcF, and RR intervals. Day -1 evening (PM) was the Baseline for participants with only Day -1 records. Day 1 PM Dose was the Baseline for participants with Day 1 records. Baseline was the mean of replicate assessments. Change from Baseline was the difference between the value at the time point analyzed and baseline value.
Time Frame: Baseline (Day 1) and up to Day 42
Population: All subjects population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: milisecond (msec)
Arm/Group | Placebo | GSK163090 1 mg | GSK163090 3 mg
Number analyzed (Participants) | 31 | 36 | 32
milisecond (msec)
  PR Interval, Day -1,PM: number analyzed (Participants) | 10 | 9 | 7
  PR Interval, Day -1,PM | 149.9 (20.06) | 148.2 (11.91) | 158.7 (16.05)
  PR Interval, Day 1PM dose,pre dose: number analyzed (Participants) | 21 | 26 | 25
  PR Interval, Day 1PM dose,pre dose | 156.4 (22.70) | 159.2 (18.43) | 163.6 (30.35)
  PR Interval, Day 2AM dose,pre dose: number analyzed (Participants) | 31 | 35 | 31
  PR Interval, Day 2AM dose,pre dose | -2.4 (9.59) | -1.2 (10.36) | -1.2 (10.01)
  PR Interval, Day 2AM dose,3 h: number analyzed (Participants) | 31 | 35 | 30
  PR Interval, Day 2AM dose,3 h | -4.1 (9.47) | -0.8 (11.12) | -3.4 (7.02)
  PR Interval, Day 2AM dose,6 h: number analyzed (Participants) | 31 | 35 | 30
  PR Interval, Day 2AM dose,6 h | -3.3 (9.14) | -2.3 (11.71) | -2.5 (7.75)
  PR Interval, Day 7AM dose,pre dose: number analyzed (Participants) | 29 | 34 | 31
  PR Interval, Day 7AM dose,pre dose | -1.5 (12.93) | -2.6 (10.99) | -1.6 (9.68)
  PR Interval, Day 7AM dose,3 h: number analyzed (Participants) | 29 | 34 | 30
  PR Interval, Day 7AM dose,3 h | -4.8 (11.71) | -1.0 (11.44) | -0.5 (8.58)
  PR Interval, Day 7AM dose,6 h: number analyzed (Participants) | 30 | 34 | 31
  PR Interval, Day 7AM dose,6 h | -1.8 (13.56) | -3.6 (11.56) | -1.8 (9.94)
  PR Interval, Day 14AM dose,pre dose: number analyzed (Participants) | 28 | 33 | 28
  PR Interval, Day 14AM dose,pre dose | 0.6 (13.78) | -1.8 (9.96) | 1.7 (9.56)
  PR Interval, Day 14AM dose,3 h: number analyzed (Participants) | 27 | 33 | 28
  PR Interval, Day 14AM dose,3 h | -3.9 (12.39) | -1.7 (11.09) | -1.4 (14.53)
  PR Interval, Day 14AM dose,6 h: number analyzed (Participants) | 28 | 33 | 28
  PR Interval, Day 14AM dose,6 h | 0.7 (11.70) | -0.8 (10.86) | -2.2 (10.00)
  PR Interval, Day 42AM dose,pre dose: number analyzed (Participants) | 25 | 25 | 24
  PR Interval, Day 42AM dose,pre dose | 1.3 (12.85) | -3.9 (10.91) | -0.2 (12.22)
  PR Interval, Day 42AM dose,3 h: number analyzed (Participants) | 25 | 25 | 24
  PR Interval, Day 42AM dose,3 h | -0.2 (14.52) | -2.9 (12.90) | -3.7 (12.85)
  PR Interval, Day 42AM dose,6 h: number analyzed (Participants) | 25 | 25 | 24
  PR Interval, Day 42AM dose,6 h | 0.3 (13.24) | -1.7 (9.20) | -2.7 (13.19)
  QRS Duration, Day -1,PM: number analyzed (Participants) | 10 | 9 | 7
  QRS Duration, Day -1,PM | 90.9 (6.90) | 86.6 (6.65) | 89.5 (5.81)
  QRS Duration, Day 1PM dose,pre dose: number analyzed (Participants) | 21 | 27 | 25
  QRS Duration, Day 1PM dose,pre dose | 90.6 (8.65) | 91.4 (8.34) | 90.0 (7.40)
  QRS Duration, Day 2AM dose,pre dose: number analyzed (Participants) | 31 | 36 | 31
  QRS Duration, Day 2AM dose,pre dose | -1.0 (6.64) | -0.6 (5.99) | -0.7 (5.59)
  QRS Duration, Day 2AM dose,3 h: number analyzed (Participants) | 31 | 36 | 31
  QRS Duration, Day 2AM dose,3 h | -0.6 (7.73) | -0.1 (6.42) | -0.1 (5.32)
  QRS Duration, Day 2AM dose,6 h: number analyzed (Participants) | 31 | 36 | 31
  QRS Duration, Day 2AM dose,6 h | -1.4 (6.82) | -0.5 (5.43) | -0.4 (5.51)
  QRS Duration, Day 7AM dose,pre dose: number analyzed (Participants) | 29 | 35 | 31
  QRS Duration, Day 7AM dose,pre dose | -1.6 (6.83) | -0.1 (5.90) | -0.3 (6.00)
  QRS Duration, Day 7AM dose,3 h: number analyzed (Participants) | 30 | 35 | 31
  QRS Duration, Day 7AM dose,3 h | -1.3 (6.67) | -1.3 (6.13) | 0.6 (5.56)
  QRS Duration, Day 7AM dose,6 h: number analyzed (Participants) | 30 | 35 | 31
  QRS Duration, Day 7AM dose,6 h | -2.0 (6.23) | -1.0 (6.77) | 0.5 (7.08)
  QRS Duration, Day 14AM dose,pre dose: number analyzed (Participants) | 28 | 34 | 28
  QRS Duration, Day 14AM dose,pre dose | -0.5 (6.90) | 0.2 (6.86) | 0.5 (6.40)
  QRS Duration, Day 14AM dose,3 h: number analyzed (Participants) | 28 | 34 | 28
  QRS Duration, Day 14AM dose,3 h | -0.4 (7.62) | -1.4 (6.32) | 1.4 (7.18)
  QRS Duration, Day 14AM dose,6 h: number analyzed (Participants) | 28 | 34 | 28
  QRS Duration, Day 14AM dose,6 h | -0.8 (7.31) | -0.3 (6.24) | 0.7 (7.57)
  QRS Duration, Day 42AM dose,pre dose: number analyzed (Participants) | 25 | 25 | 24
  QRS Duration, Day 42AM dose,pre dose | -0.5 (8.67) | -0.4 (5.65) | -1.0 (6.75)
  QRS Duration, Day 42AM dose,3 h: number analyzed (Participants) | 25 | 25 | 24
  QRS Duration, Day 42AM dose,3 h | 0.0 (8.55) | -0.9 (5.50) | 0.3 (6.12)
  QRS Duration, Day 42AM dose,6 h: number analyzed (Participants) | 25 | 25 | 24
  QRS Duration, Day 42AM dose,6 h | 0.5 (8.56) | 0.6 (5.87) | 1.2 (6.63)
  QT Interval, Day -1,PM: number analyzed (Participants) | 10 | 9 | 7
  QT Interval, Day -1,PM | 390.4 (19.42) | 375.1 (31.50) | 377.3 (30.89)
  QT Interval, Day 1PM dose,pre dose: number analyzed (Participants) | 21 | 26 | 25
  QT Interval, Day 1PM dose,pre dose | 372.4 (22.92) | 382.2 (16.07) | 380.7 (24.77)
  QT Interval, Day 2AM dose,pre dose: number analyzed (Participants) | 31 | 35 | 30
  QT Interval, Day 2AM dose,pre dose | -2.0 (24.13) | -3.2 (26.99) | -2.6 (20.37)
  QT Interval, Day 2AM dose,3 h: number analyzed (Participants) | 31 | 34 | 30
  QT Interval, Day 2AM dose,3 h | -7.7 (21.57) | -3.8 (28.15) | -7.0 (21.73)
  QT Interval, Day 2AM dose,6 h: number analyzed (Participants) | 31 | 34 | 30
  QT Interval, Day 2AM dose,6 h | -4.7 (21.43) | -6.1 (27.41) | -7.5 (17.92)
  QT Interval, Day 7AM dose,pre dose: number analyzed (Participants) | 29 | 33 | 30
  QT Interval, Day 7AM dose,pre dose | 1.3 (21.92) | -2.8 (19.98) | -0.0 (22.90)
  QT Interval, Day 7AM dose,3 h: number analyzed (Participants) | 29 | 34 | 30
  QT Interval, Day 7AM dose,3 h | -3.7 (23.26) | -2.7 (18.10) | -1.7 (21.36)
  QT Interval, Day 7AM dose,6 h: number analyzed (Participants) | 30 | 34 | 31
  QT Interval, Day 7AM dose,6 h | -4.6 (20.57) | -6.0 (19.66) | -1.9 (21.24)
  QT Interval, Day 14AM dose,pre dose: number analyzed (Participants) | 28 | 32 | 28
  QT Interval, Day 14AM dose,pre dose | 5.9 (22.87) | 2.7 (14.97) | 0.3 (23.61)
  QT Interval, Day 14AM dose,3 h: number analyzed (Participants) | 28 | 33 | 28
  QT Interval, Day 14AM dose,3 h | -1.6 (23.64) | -5.0 (20.32) | -3.0 (23.36)
  QT Interval, Day 14AM dose,6 h | 0.2 (21.32) | -5.0 (19.46) | 0.3 (21.26)
  QT Interval, Day 42AM dose,pre dose: number analyzed (Participants) | 25 | 25 | 23
  QT Interval, Day 42AM dose,pre dose | 5.5 (25.30) | -1.6 (29.31) | 4.1 (23.30)
  QT Interval, Day 42AM dose,3 h: number analyzed (Participants) | 25 | 25 | 24
  QT Interval, Day 42AM dose,3 h | -0.2 (22.81) | -2.4 (26.68) | -2.0 (24.82)
  QT Interval, Day 42AM dose,6 h: number analyzed (Participants) | 25 | 25 | 24
  QT Interval, Day 42AM dose,6 h | 3.4 (24.63) | -2.6 (30.94) | -3.7 (23.97)
  QTcB, Day -1,PM: number analyzed (Participants) | 10 | 9 | 7
  QTcB, Day -1,PM | 428.5 (14.64) | 422.6 (25.22) | 410.5 (17.28)
  QTcB, Day 1PM dose,pre dose: number analyzed (Participants) | 21 | 26 | 25
  QTcB, Day 1PM dose,pre dose | 418.6 (21.11) | 417.5 (18.51) | 419.3 (19.28)
  QTcB, Day 2AM dose,pre dose: number analyzed (Participants) | 31 | 35 | 30
  QTcB, Day 2AM dose,pre dose | -3.8 (13.48) | 1.6 (18.90) | -2.6 (14.77)
  QTcB, Day 2AM dose,3 h: number analyzed (Participants) | 31 | 34 | 30
  QTcB, Day 2AM dose,3 h | -7.7 (15.30) | -1.1 (17.44) | -0.9 (14.65)
  QTcB, Day 2AM dose,6 h: number analyzed (Participants) | 31 | 34 | 30
  QTcB, Day 2AM dose,6 h | -5.5 (16.93) | -1.6 (18.49) | -0.2 (13.68)
  QTcB, Day 7AM dose,pre dose: number analyzed (Participants) | 29 | 33 | 30
  QTcB, Day 7AM dose,pre dose | -2.2 (17.77) | -3.9 (22.66) | 3.6 (13.96)
  QTcB, Day 7AM dose,3 h: number analyzed (Participants) | 29 | 34 | 30
  QTcB, Day 7AM dose,3 h | -6.4 (19.71) | -2.4 (20.53) | 1.9 (18.00)
  QTcB, Day 7AM dose,6 h: number analyzed (Participants) | 30 | 34 | 31
  QTcB, Day 7AM dose,6 h | -4.3 (16.62) | -2.9 (19.49) | 4.3 (16.82)
  QTcF, Day -1,PM: number analyzed (Participants) | 10 | 9 | 7
  QTcF, Day -1,PM | 415.30 (12.440) | 405.66 (17.954) | 398.97 (20.232)
  QTcF, Day 1PM dose,pre dose: number analyzed (Participants) | 21 | 26 | 25
  QTcF, Day 1PM dose,pre dose | 402.47 (18.503) | 405.24 (12.952) | 405.76 (14.431)
  QTcF, Day 2AM dose,pre dose: number analyzed (Participants) | 31 | 35 | 30
  QTcF, Day 2AM dose,pre dose | -3.28 (15.070) | -0.05 (18.340) | -2.70 (13.592)
  QTcF, Day 2AM dose,3 h: number analyzed (Participants) | 31 | 34 | 30
  QTcF, Day 2AM dose,3 h | -7.78 (14.789) | -2.22 (18.127) | -3.10 (11.385)
  QTcF, Day 2AM dose,6 h: number analyzed (Participants) | 31 | 34 | 30
  QTcF, Day 2AM dose,6 h | -5.28 (15.945) | -3.29 (17.988) | -2.80 (8.543)
  QTcF, Day 7AM dose,pre dose: number analyzed (Participants) | 29 | 33 | 30
  QTcF, Day 7AM dose,pre dose | -1.03 (15.456) | -3.59 (17.264) | 2.43 (10.501)
  QTcF, Day 7AM dose,3 h: number analyzed (Participants) | 29 | 34 | 30
  QTcF, Day 7AM dose,3 h | -5.47 (16.491) | -2.59 (14.017) | 0.70 (12.787)
  QTcF, Day 7AM dose,6 h: number analyzed (Participants) | 30 | 34 | 31
  QTcF, Day 7AM dose,6 h | -4.47 (14.499) | -4.08 (14.692) | 2.18 (12.292)
  QTcF, Day 14AM dose,pre dose: number analyzed (Participants) | 28 | 32 | 28
  QTcF, Day 14AM dose,pre dose | -1.44 (16.241) | -0.26 (15.470) | 0.60 (12.221)
  QTcF, Day 14AM dose,3 h: number analyzed (Participants) | 28 | 33 | 28
  QTcF, Day 14AM dose,3 h | -2.15 (14.577) | -4.21 (14.874) | -0.70 (16.000)
  QTcF, Day 14AM dose,6 h: number analyzed (Participants) | 28 | 33 | 28
  QTcF, Day 14AM dose,6 h | -2.40 (14.801) | -3.72 (15.555) | 3.02 (12.372)
  QTcF, Day 42AM dose,pre dose: number analyzed (Participants) | 25 | 25 | 23
  QTcF, Day 42AM dose,pre dose | -1.10 (14.014) | 0.28 (18.937) | 6.02 (11.852)
  QTcF, Day 42AM dose,3 h: number analyzed (Participants) | 25 | 25 | 24
  QTcF, Day 42AM dose,3 h | -4.24 (14.575) | -1.68 (15.447) | 1.76 (12.233)
  QTcF, Day 42AM dose,6 h: number analyzed (Participants) | 25 | 25 | 24
  QTcF, Day 42AM dose,6 h | -1.58 (15.354) | -0.32 (18.769) | 1.50 (16.181)
  RR Interval, Day -1,PM: number analyzed (Participants) | 10 | 9 | 7
  RR Interval, Day -1,PM | 833.92 (94.941) | 803.45 (179.989) | 848.28 (101.842)
  RR Interval, Day 1PM dose,pre dose: number analyzed (Participants) | 21 | 26 | 25
  RR Interval, Day 1PM dose,pre dose | 796.78 (100.400) | 844.79 (105.834) | 834.03 (146.780)
  RR Interval, Day 2AM dose,pre dose: number analyzed (Participants) | 31 | 35 | 30
  RR Interval, Day 2AM dose,pre dose | 8.52 (87.037) | -22.39 (110.999) | 1.77 (92.320)
  RR Interval, Day 2AM dose,3 h: number analyzed (Participants) | 31 | 34 | 30
  RR Interval, Day 2AM dose,3 h | -0.62 (90.126) | -12.00 (115.655) | -26.77 (131.444)
  RR Interval, Day 2AM dose,6 h: number analyzed (Participants) | 31 | 34 | 30
  RR Interval, Day 2AM dose,6 h | 2.50 (84.105) | -20.53 (117.183) | -31.09 (124.683)
  RR Interval, Day 7AM dose,pre dose: number analyzed (Participants) | 29 | 33 | 30
  RR Interval, Day 7AM dose,pre dose | 16.29 (105.628) | 5.20 (122.749) | -17.08 (127.229)
  RR Interval, Day 7AM dose,3 h: number analyzed (Participants) | 29 | 34 | 30
  RR Interval, Day 7AM dose,3 h | 10.29 (115.521) | -0.40 (119.174) | -17.24 (128.785)
  RR Interval, Day 7AM dose,6 h: number analyzed (Participants) | 30 | 34 | 31
  RR Interval, Day 7AM dose,6 h | -2.24 (97.793) | -14.65 (122.435) | -27.36 (125.990)
  RR Interval, Day 14AM dose,pre dose: number analyzed (Participants) | 28 | 32 | 28
  RR Interval, Day 14AM dose,pre dose | 52.74 (140.757) | 20.29 (106.077) | -4.41 (109.804)
  RR Interval, Day 14AM dose,3 h: number analyzed (Participants) | 28 | 33 | 28
  RR Interval, Day 14AM dose,3 h | 3.28 (122.146) | -8.39 (116.181) | -17.71 (112.985)
  RR Interval, Day 14AM dose,6 h: number analyzed (Participants) | 28 | 33 | 28
  RR Interval, Day 14AM dose,6 h | 17.25 (103.448) | -8.28 (120.157) | -18.59 (108.155)
  RR Interval, Day 42AM dose,pre dose: number analyzed (Participants) | 25 | 25 | 23
  RR Interval, Day 42AM dose,pre dose | 46.40 (126.076) | -13.44 (145.953) | -11.87 (125.389)
  RR Interval, Day 42AM dose,3 h: number analyzed (Participants) | 25 | 25 | 24
  RR Interval, Day 42AM dose,3 h | 28.22 (111.532) | -6.81 (148.104) | -26.69 (127.058)
  RR Interval, Day 42AM dose,6 h: number analyzed (Participants) | 25 | 25 | 24
  RR Interval, Day 42AM dose,6 h | 35.60 (124.148) | -17.57 (167.309) | -35.87 (132.117)

11. Primary Outcome: Mean of Change From Baseline in Systolic and Diastolic Blood Pressure (BP)
Description: Semi-supine systolic and diastolic blood pressure was assessed at the specified time points. Measurements were taken after the participant has been semi-supine for at least 5 minutes. BP was measured at least every hour until the values were within the normal range. Day 1 was Baseline and change from Baseline was difference between the value at the time point analyzed and baseline value.
Time Frame: Baseline (Day 1) , Day 2, 3, 4, 5, 6, 7, 8, 14, 21, 28 and 42
Population: All subjects population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo | GSK163090 1 mg | GSK163090 3 mg
Number analyzed (Participants) | 31 | 36 | 32
Millimeters of mercury (mmHg)
  Systolic BP, Day 1PM dose,pre dose: number analyzed (Participants) | 30 | 36 | 32
  Systolic BP, Day 1PM dose,pre dose | 120.6 (10.65) | 120.3 (9.31) | 120.9 (13.84)
  Systolic BP, Day 1PM dose,2 h | -0.8 (3.55) | 0.1 (4.53) | 1.5 (8.16)
  Systolic BP ,Day 2AM dose,pre dose: number analyzed (Participants) | 31 | 36 | 31
  Systolic BP ,Day 2AM dose,pre dose | -0.8 (5.19) | 1.2 (5.98) | 1.0 (5.55)
  Systolic BP ,Day 2AM dose,3 h: number analyzed (Participants) | 31 | 36 | 31
  Systolic BP ,Day 2AM dose,3 h | -0.1 (4.33) | 1.0 (5.51) | 1.1 (6.53)
  Systolic BP ,Day 2AM dose,6 h: number analyzed (Participants) | 31 | 36 | 31
  Systolic BP ,Day 2AM dose,6 h | -1.2 (3.80) | 0.2 (4.34) | 2.1 (8.53)
  Systolic BP ,Day 2PM dose,1 h: number analyzed (Participants) | 31 | 36 | 31
  Systolic BP ,Day 2PM dose,1 h | -0.5 (4.42) | 0.3 (4.80) | 0.4 (8.35)
  Systolic BP ,Day 3AM dose,pre dose: number analyzed (Participants) | 31 | 36 | 31
  Systolic BP ,Day 3AM dose,pre dose | -1.6 (9.23) | 0.4 (5.84) | -1.1 (6.01)
  Systolic BP ,Day 3AM dose,3 h: number analyzed (Participants) | 31 | 36 | 31
  Systolic BP ,Day 3AM dose,3 h | -1.2 (6.98) | 0.5 (7.10) | -0.8 (5.32)
  Systolic BP ,Day 4AM dose,pre dose: number analyzed (Participants) | 31 | 36 | 31
  Systolic BP ,Day 4AM dose,pre dose | -0.1 (5.44) | -0.2 (5.19) | -0.2 (6.07)
  Systolic BP ,Day 4AM dose,3 h: number analyzed (Participants) | 30 | 36 | 31
  Systolic BP ,Day 4AM dose,3 h | 0.5 (5.02) | 2.1 (7.07) | -0.3 (5.22)
  Systolic BP ,Day 5AM dose,pre dose: number analyzed (Participants) | 31 | 35 | 31
  Systolic BP ,Day 5AM dose,pre dose | -1.4 (5.97) | -0.7 (5.16) | 0.5 (6.72)
  Systolic BP ,Day 5AM dose,3 h: number analyzed (Participants) | 31 | 35 | 31
  Systolic BP ,Day 5AM dose,3 h | -0.8 (4.43) | -0.8 (5.18) | -0.6 (4.97)
  Systolic BP ,Day 6AM dose,pre dose: number analyzed (Participants) | 31 | 35 | 31
  Systolic BP ,Day 6AM dose,pre dose | -2.9 (5.19) | -0.2 (6.01) | 0.6 (7.08)
  Systolic BP ,Day 6AM dose,3 h: number analyzed (Participants) | 31 | 35 | 31
  Systolic BP ,Day 6AM dose,3 h | 0.2 (4.48) | 0.5 (5.72) | 1.7 (8.65)
  Systolic BP ,Day 7AM dose,pre dose: number analyzed (Participants) | 30 | 35 | 31
  Systolic BP ,Day 7AM dose,pre dose | -1.4 (6.98) | 0.8 (6.65) | 2.8 (8.24)
  Systolic BP ,Day 7AM dose,3 h: number analyzed (Participants) | 30 | 35 | 31
  Systolic BP ,Day 7AM dose,3 h | -0.8 (6.39) | 0.1 (7.42) | 2.7 (5.70)
  Systolic BP ,Day 7AM dose,6 h: number analyzed (Participants) | 30 | 35 | 31
  Systolic BP ,Day 7AM dose,6 h | 1.5 (5.77) | 0.2 (5.29) | 2.8 (6.97)
  Systolic BP ,Day 7PM dose,1h: number analyzed (Participants) | 30 | 35 | 31
  Systolic BP ,Day 7PM dose,1h | -0.2 (6.11) | -0.7 (7.78) | 2.1 (9.20)
  Systolic BP ,Day 8AM dose,pre dose: number analyzed (Participants) | 29 | 35 | 30
  Systolic BP ,Day 8AM dose,pre dose | -1.8 (5.18) | -0.3 (8.34) | 0.3 (6.96)
  Systolic BP ,Day 8AM dose,3 h: number analyzed (Participants) | 29 | 35 | 30
  Systolic BP ,Day 8AM dose,3 h | -1.0 (6.02) | -0.6 (6.94) | 1.4 (7.25)
  Systolic BP ,Day 14AM dose,pre dose: number analyzed (Participants) | 28 | 34 | 29
  Systolic BP ,Day 14AM dose,pre dose | -3.0 (6.77) | 1.0 (5.71) | 0.3 (8.16)
  Systolic BP ,Day 14AM dose,3 h: number analyzed (Participants) | 28 | 34 | 28
  Systolic BP ,Day 14AM dose,3 h | -0.8 (7.65) | 0.9 (7.82) | 1.6 (8.00)
  Systolic BP ,Day 14AM dose,6 h: number analyzed (Participants) | 28 | 34 | 28
  Systolic BP ,Day 14AM dose,6 h | -1.1 (8.03) | 1.6 (8.10) | 1.3 (8.86)
  Systolic BP ,Day 14PM dose,1h: number analyzed (Participants) | 28 | 34 | 28
  Systolic BP ,Day 14PM dose,1h | -2.0 (6.98) | 0.3 (7.48) | 1.8 (9.86)
  Systolic BP ,Day 21AM dose,pre dose: number analyzed (Participants) | 28 | 30 | 28
  Systolic BP ,Day 21AM dose,pre dose | -1.8 (6.73) | 0.0 (6.99) | 0.5 (8.43)
  Systolic BP ,Day 21AM dose,3 h: number analyzed (Participants) | 28 | 30 | 28
  Systolic BP ,Day 21AM dose,3 h | -2.1 (7.20) | 0.7 (7.34) | 1.5 (10.43)
  Systolic BP ,Day 28AM dose,pre dose: number analyzed (Participants) | 27 | 26 | 27
  Systolic BP ,Day 28AM dose,pre dose | -1.4 (7.36) | -1.6 (5.95) | 2.9 (7.59)
  Systolic BP ,Day 28AM dose,3 h: number analyzed (Participants) | 27 | 26 | 27
  Systolic BP ,Day 28AM dose,3 h | -1.2 (6.38) | 1.9 (6.23) | 3.2 (8.32)
  Systolic BP ,Day 42AM dose,pre dose: number analyzed (Participants) | 25 | 25 | 24
  Systolic BP ,Day 42AM dose,pre dose | 0.1 (6.71) | 1.1 (6.95) | 0.3 (7.71)
  Systolic BP ,Day 42AM dose,3 h: number analyzed (Participants) | 25 | 25 | 24
  Systolic BP ,Day 42AM dose,3 h | -1.8 (6.32) | 2.7 (5.91) | 2.0 (9.17)
  Diastolic BP, Day 1PM dose,pre dose: number analyzed (Participants) | 30 | 36 | 32
  Diastolic BP, Day 1PM dose,pre dose | 76.2 (5.83) | 75.6 (5.95) | 76.8 (7.91)
  Diastolic BP, Day 1PM dose,2 h | -0.4 (3.53) | 0.4 (3.30) | 0.7 (5.24)
  Diastolic BP ,Day 2AM dose,pre dose | -0.7 (2.93) | -0.0 (3.65) | -0.2 (5.67)
  Diastolic BP ,Day 2AM dose,3 h | -1.2 (2.88) | 0.7 (4.85) | 0.1 (4.03)
  Diastolic BP ,Day 2AM dose,6 h | -0.8 (4.56) | -0.3 (3.88) | 1.3 (5.51)
  Diastolic BP ,Day 2PM dose,1 h | 0.1 (3.83) | -0.0 (4.19) | -0.4 (6.45)
  Diastolic BP ,Day 3AM dose,pre dose | -2.5 (4.41) | -0.1 (4.41) | -0.9 (6.53)
  Diastolic BP ,Day 3AM dose,3 h | -2.3 (4.68) | 0.3 (4.87) | -0.4 (5.68)
  Diastolic BP ,Day 4AM dose,pre dose | -1.9 (4.93) | 0.2 (4.35) | -0.7 (4.56)
  Diastolic Systolic BP ,Day 4AM dose,3 h | -2.6 (5.15) | 0.0 (6.50) | -1.4 (4.85)
  Diastolic BP ,Day 5AM dose,pre dose | -1.9 (4.94) | 0.4 (4.17) | -1.9 (5.42)
  Diastolic BP ,Day 5AM dose,3 h | -1.2 (3.99) | -0.2 (4.04) | -1.7 (4.88)
  Diastolic BP ,Day 6AM dose,pre dose | -1.3 (4.68) | 0.2 (5.06) | -1.7 (6.45)
  Diastolic BP ,Day 6AM dose,3 h | -1.8 (5.29) | -0.2 (5.01) | -1.2 (7.14)
  Diastolic BP ,Day 7AM dose,pre dose | -2.1 (5.87) | 0.1 (7.66) | 0.3 (6.67)
  Diastolic BP ,Day 7AM dose,3 h | -1.2 (5.56) | -0.1 (6.19) | -0.6 (5.56)
  Diastolic BP ,Day 7AM dose,6 h | -1.0 (4.16) | -0.7 (4.27) | -0.6 (5.75)
  Diastolic BP ,Day 7PM dose,1h | -1.5 (4.21) | -0.3 (5.17) | -0.9 (7.12)
  Diastolic BP ,Day 8AM dose,pre dose | -1.7 (5.36) | -0.5 (6.81) | -1.9 (7.14)
  Diastolic BP ,Day 8AM dose,3 h | -1.7 (5.62) | -0.6 (6.18) | -0.7 (7.83)
  Diastolic BP ,Day 14AM dose,pre dose | -2.7 (5.34) | -1.0 (5.57) | -0.2 (7.61)
  Diastolic BP ,Day 14AM dose,3 h | -2.2 (5.11) | 0.0 (6.84) | -0.6 (7.21)
  Diastolic BP ,Day 14AM dose,6 h | -2.8 (5.60) | 0.1 (6.54) | -0.8 (6.39)
  Diastolic BP ,Day 14PM dose,1h | -2.8 (5.14) | -0.3 (5.03) | -0.9 (6.69)
  Diastolic BP ,Day 21AM dose,pre dose | -2.9 (5.10) | 0.5 (5.38) | -0.8 (7.63)
  Diastolic BP ,Day 21AM dose,3 h | -2.7 (5.35) | -0.8 (5.82) | -1.7 (7.43)
  Diastolic BP ,Day 28AM dose,pre dose | -2.0 (5.12) | -0.9 (4.44) | 0.1 (6.72)
  Diastolic BP ,Day 28AM dose,3 h | -2.1 (5.09) | 1.4 (4.50) | -1.4 (6.40)
  Diastolic BP ,Day 42AM dose,pre dose | 0.4 (7.37) | 0.7 (5.25) | -0.2 (7.57)
  Diastolic BP ,Day 42AM dose,3 h | -1.7 (7.39) | 2.5 (4.70) | -0.6 (7.66)

12. Primary Outcome: Mean of Change From Baseline in Heart Rate
Description: Heart rate is the speed of the heartbeat measured by the number of contractions of the heart per minute, (beats per minute). Heart rate was assessed at the specified time points. Measurements were taken after the participant has been semi-supine for at least 5 minutes. Day 1 was Baseline and change from Baseline was difference between the value at the time point analyzed and baseline value.
Time Frame: Baseline (Day 1), Day 2, 3, 4, 5, 6, 7, 8, 14, 21, 28 and 42
Population: All subjects population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GSK163090 1 mg | GSK163090 3 mg
Number analyzed (Participants) | 31 | 36 | 32
Beats per minute
  Heart rate, Day 1PM dose,pre dose: number analyzed (Participants) | 30 | 36 | 32
  Heart rate, Day 1PM dose,pre dose | 73.0 (7.54) | 73.3 (10.67) | 71.8 (7.43)
  Heart rate, Day 1PM dose,2 h | 1.4 (6.83) | 1.0 (4.63) | 1.1 (5.12)
  Heart rate,Day 2AM dose,pre dose: number analyzed (Participants) | 31 | 36 | 31
  Heart rate,Day 2AM dose,pre dose | -0.8 (5.73) | 0.4 (8.27) | 1.3 (6.63)
  Heart rate,Day 2AM dose,3 h: number analyzed (Participants) | 31 | 36 | 31
  Heart rate,Day 2AM dose,3 h | 0.8 (5.19) | 0.8 (7.99) | 2.5 (6.47)
  Heart rate,Day 2AM dose,6 h: number analyzed (Participants) | 31 | 36 | 31
  Heart rate,Day 2AM dose,6 h | 0.2 (6.08) | 1.9 (7.27) | 2.8 (6.56)
  Heart rate,Day 2PM dose,1 h: number analyzed (Participants) | 31 | 36 | 31
  Heart rate,Day 2PM dose,1 h | 0.6 (7.02) | 1.0 (6.72) | 2.4 (7.28)
  Heart rate,Day 3AM dose,pre dose: number analyzed (Participants) | 31 | 36 | 31
  Heart rate,Day 3AM dose,pre dose | -0.7 (8.49) | 1.2 (6.49) | 1.3 (6.85)
  Heart rate,Day 3AM dose,3 h: number analyzed (Participants) | 31 | 36 | 31
  Heart rate,Day 3AM dose,3 h | 0.1 (8.26) | 2.6 (6.70) | 2.0 (5.38)
  Heart rate,Day 4AM dose,pre dose: number analyzed (Participants) | 31 | 36 | 31
  Heart rate,Day 4AM dose,pre dose | -0.3 (10.04) | 0.7 (7.15) | 1.2 (5.03)
  Heart rate,Day 4AM dose,3 h: number analyzed (Participants) | 30 | 36 | 31
  Heart rate,Day 4AM dose,3 h | 0.9 (8.23) | 1.7 (7.82) | 1.3 (5.65)
  Heart rate,Day 5AM dose,pre dose: number analyzed (Participants) | 31 | 35 | 31
  Heart rate,Day 5AM dose,pre dose | -0.4 (7.48) | -0.5 (6.48) | 1.0 (6.36)
  Heart rate,Day 5AM dose,3 h: number analyzed (Participants) | 31 | 35 | 31
  Heart rate,Day 5AM dose,3 h | 0.1 (8.54) | 0.6 (6.09) | 1.7 (5.87)
  Heart rate,Day 6AM dose,pre dose: number analyzed (Participants) | 31 | 35 | 31
  Heart rate,Day 6AM dose,pre dose | 1.7 (10.54) | 0.2 (6.87) | 0.8 (5.43)
  Heart rate,Day 6AM dose,3 h: number analyzed (Participants) | 31 | 35 | 31
  Heart rate,Day 6AM dose,3 h | 0.2 (9.42) | 0.4 (7.01) | -0.3 (7.60)
  Heart rate,Day 7AM dose,pre dose: number analyzed (Participants) | 30 | 35 | 31
  Heart rate,Day 7AM dose,pre dose | -0.8 (9.79) | -1.0 (6.95) | 2.4 (6.51)
  Heart rate,Day 7AM dose,3 h: number analyzed (Participants) | 30 | 35 | 31
  Heart rate,Day 7AM dose,3 h | -0.7 (8.74) | -0.1 (6.94) | 2.1 (6.76)
  Heart rate,Day 7AM dose,6 h: number analyzed (Participants) | 30 | 35 | 31
  Heart rate,Day 7AM dose,6 h | -1.3 (9.81) | -0.4 (7.67) | 3.0 (7.08)
  Heart rate,Day 7PM dose,1h: number analyzed (Participants) | 30 | 35 | 31
  Heart rate,Day 7PM dose,1h | -0.6 (9.83) | 0.2 (7.21) | 2.5 (6.64)
  Heart rate BP ,Day 8AM dose,pre dose: number analyzed (Participants) | 29 | 35 | 30
  Heart rate BP ,Day 8AM dose,pre dose | -0.7 (8.38) | -0.4 (7.55) | 1.5 (5.98)
  Heart rate,Day 8AM dose,3 h: number analyzed (Participants) | 29 | 35 | 30
  Heart rate,Day 8AM dose,3 h | -0.7 (8.55) | 0.2 (6.31) | 1.7 (5.60)
  Heart rate,Day 14AM dose,pre dose: number analyzed (Participants) | 28 | 34 | 29
  Heart rate,Day 14AM dose,pre dose | -2.1 (11.59) | 0.3 (6.37) | -0.5 (6.09)
  Heart rate,Day 14AM dose,3 h: number analyzed (Participants) | 28 | 34 | 28
  Heart rate,Day 14AM dose,3 h | 1.2 (10.56) | 2.5 (6.26) | 0.6 (5.51)
  Heart rate,Day 14AM dose,6 h: number analyzed (Participants) | 28 | 34 | 28
  Heart rate,Day 14AM dose,6 h | 1.6 (11.28) | 2.3 (6.60) | 0.7 (6.13)
  Heart rate,Day 14PM dose,1h | -0.8 (9.40) | 0.6 (6.36) | 0.4 (5.49)
  Heart rate,Day 21AM dose,pre dose: number analyzed (Participants) | 28 | 30 | 28
  Heart rate,Day 21AM dose,pre dose | -0.3 (9.36) | -0.3 (7.70) | 2.4 (6.54)
  Heart rate,Day 21AM dose,3 h: number analyzed (Participants) | 28 | 30 | 28
  Heart rate,Day 21AM dose,3 h | -0.5 (9.17) | 1.2 (6.99) | 2.1 (6.57)
  Heart rate,Day 28AM dose,pre dose: number analyzed (Participants) | 27 | 26 | 27
  Heart rate,Day 28AM dose,pre dose | -1.6 (8.44) | -0.8 (7.64) | 1.3 (5.97)
  Heart rate,Day 28AM dose,3 h: number analyzed (Participants) | 27 | 26 | 27
  Heart rate,Day 28AM dose,3 h | -0.7 (8.92) | -0.3 (6.28) | 2.4 (6.28)
  Heart rate,Day 42AM dose,pre dose: number analyzed (Participants) | 25 | 25 | 24
  Heart rate,Day 42AM dose,pre dose | -2.4 (11.05) | -0.8 (7.13) | 1.1 (5.89)
  Heart rate,Day 42AM dose,3 h: number analyzed (Participants) | 25 | 25 | 24
  Heart rate,Day 42AM dose,3 h | -1.4 (9.69) | -0.6 (8.33) | 1.3 (7.38)

13. Primary Outcome: Number of Participants With All Adverse Events (AEs), and Serious Adverse Events (SAEs)
Description: Data for number of participants who presented one or more adverse events (serious or non serious) was reported. An AE was defined as any untoward medical occurrence (MO) in a participant temporally associated with the use of a medicinal product (MP), whether or not considered related to the MP and can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with its use. The SAE was any untoward MO that, at any dose, results in death, life threatening, persistent or significant disability/incapacity, results in or prolongs inpatient hospitalization, congenital abnormality or birth defect, that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition.
Time Frame: Up to Day 52
Population: All subjects population. The number of participants available at the particular time point were used for analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK163090 1 mg | GSK163090 3 mg
Number analyzed (Participants) | 31 | 36 | 32
Participants
  Any AE | 17 | 24 | 14
  Any SAE | 0 | 0 | 0

14. Secondary Outcome: Mean Last Observed Quantifiable Concentration (Ct) of GSK163090 Over the Period
Description: Ctrough is defined as trough plasma concentration (measured concentration at the end of a dosing interval at steady state [taken directly before next administration]). Concentration was reported at specified time points.
Time Frame: Day 4 (AM pre-dose), Day 7 (AM and PM pre-dose), Day 10 (AM and PM pre-dose), Day 14 (AM and PM pre-dose), Day 21 (AM pre dose), Day 28 (AM pre dose), Day 42 (AM pre-dose and 4-6 h post AM dose)
Population: The 'PK population' comprised of participants in the intent to treat population for whom a pharmacokinetic sample was obtained and analyzed.
Measure: Mean (Standard Deviation); unit: microgram per liter
Arm/Group | GSK163090 1 mg | GSK163090 3 mg
Number analyzed (Participants) | 285 | 247
microgram per liter | 0.951 (0.6987) | 3.239 (2.1849)

15. Secondary Outcome: Area Under Concentration-time Curve (AUC) at Steady State
Description: PK samples were supposed to be collected to estimate individual specific parameters like AUC however data for this outcome was not collected.
Time Frame: as for outcome 14
Population: PK population.
Arm/Group | GSK163090 1 mg | GSK163090 3 mg
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Average Concentration (Cave) at Steady State
Description: PK samples were supposed to be collected to estimate individual specific parameters like Cave however data for this outcome was not collected.
Time Frame: as for outcome 14
Population: PK population.
Arm/Group | GSK163090 1 mg | GSK163090 3 mg
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Preliminary Pharmacokinetic/ Pharmacodynamic (PK/PD)Relationships for GSK163090 in Participants With MDD.
Description: PK/PD relationships for GSK163090 in participants with MDD data was not collected.
Time Frame: as for outcome 14
Population: PK population.
Arm/Group | GSK163090 1 mg | GSK163090 3 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 52
Description: All Subjects population was used.
Groups:
- GSK163090 1 mg: Participants were randomized to the low dose arm to receive oral dose of GSK163090 up to 1 mg immediate release tablet twice a day, with one tablet in the AM and one taken between 11 to 13 hours after the AM dose in the PM for 6 weeks. Daily dosage was provided according to the titration schedule, where the participants received (AM -matching placebo tablet, PM- GSK163090 0.5 mg ) on Day 1 and continued (AM- GSK163090 0.5 mg and PM- GSK163090 0.5 mg).from Day 2 onwards.
Arm/Group | Placebo | GSK163090 1 mg | GSK163090 3 mg
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/36 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/36 | 0/32
Other Adverse Events (participants affected / at risk) | 17/31 | 24/36 | 14/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=31) | GSK163090 1 mg (N=36) | GSK163090 3 mg (N=32)
Headache (Nervous system disorders) | 4 | 5 | 4
Dizziness (Nervous system disorders) | 2 | 4 | 2
Somnolence (Nervous system disorders) | 1 | 3 | 0
Akathisia (Nervous system disorders) | 0 | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 1
Psychomotor hyperactivity (Nervous system disorders) | 0 | 1 | 1
Mental retardation (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 4 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 3 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 0
Blood pressure increased (Investigations) | 0 | 2 | 0
Thyroxine decreased (Investigations) | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 1
Blood urea increased (Investigations) | 1 | 0 | 0
CSF test abnormal (Investigations) | 0 | 1 | 0
Carbohydrate tolerance decreased (Investigations) | 0 | 0 | 1
Electrocardiogram PR shortened (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
Protein urine (Investigations) | 0 | 1 | 0
Urine ketone body present (Investigations) | 0 | 1 | 0
Urine leukocyte esterase (Investigations) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 1 | 4
Insomnia (Psychiatric disorders) | 1 | 3 | 3
Depression (Psychiatric disorders) | 1 | 1 | 1
Agitation (Psychiatric disorders) | 1 | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 4 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 2 | 1
Tachycardia (Cardiac disorders) | 0 | 2 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 1
Irritability (General disorders) | 0 | 1 | 0
Sensation of foreign body (General disorders) | 0 | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0
Enuresis (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.